CLINICAL TRIAL: NCT00182832
Title: Enhancing Care for Hospitalized Older Adults With Cognitive Impairment
Brief Title: e-CHAMP: Enhancing Care for Hospitalized Older Adults With Memory Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Malaz Boustani, MD, MPH, Principal Investigator, Regenstrief Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IA0077; K23AG026770 (NIH); K23AG026779-01
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Cognitive Impairment; Delirium
Keywords: Physician Behavior; Hospital Acquired Complications; MCI; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Delirium | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: e-CHAMP (Enhancing Care for Hospitalized Older Adults with Cognitive Impairment)
- 2 (Active Comparator)
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: e-CHAMP (Enhancing Care for Hospitalized Older Adults with Cognitive Impairment) — Cognitive screening plus Computerized Decision Support System: proactive screening program for cognitive impairment combined with computerized review of the electronic medical record
  Other Names: CDSS
  Arms: 1
Behavioral: Standard Care — Standard care for hospitalized older patients with cognitive impairment
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a cognitive screening program coupled with a computerized decision support system in improving the quality of care for hospitalized older adults with cognitive impairment.

DETAILED DESCRIPTION:
A growing body of evidence demonstrates that older patients with cognitive impairment (CI) who are hospitalized for the management of their medical illnesses are especially vulnerable to hospital acquired complications such as falls, injuries, pressure ulcers, restraints, and delirium. These complications contribute to mortality, poorer functional status, limited rehabilitation, prolonged length of stay, increased institutionalization, and higher health care costs. Evidence suggests that interdisciplinary geriatric inpatient services improve care for hospitalized older adults without CI; however, their effectiveness among older adults with CI is less clear. One reason may be the ever-quickening pace of care in the hospital setting. Thus, matching geriatric evaluation and recommendations to the true pace of hospital care may be one mechanism to improve the care of older adults with CI.

A recent report from the Institute of Medicine suggested that integrating information technology (IT) into health care is the best route to improve the overall safety and quality of the health care system. The hypothesis of this study is that missed, delayed, post-hoc, and incomplete implementation of the geriatric service-based recommendations are significant factors explaining the poor outcomes among hospitalized older adults with cognitive impairment (CI). Wishard Memorial Hospital's physicians are already using a Computerized Decision Support System (CDSS), developed by the Regenstrief Institute, to guide their medical services. For this study, the content of this CDSS will be modified to the special needs of older adults with CI. A major advantage of such a system is reducing the time to implementation of geriatric recommendations with a specific focus on preventing the initiation of potentially harmful medications and procedures during the critical first 48 hours of hospitalization.

A total of 400 patients with cognitive impairment who have been hospitalized in a medical ward will be recruited for this study. Patients will be randomized to receive either standard care or the proactive screening program for CI combined with the modified CDSS. The electronic medical record for all patients will be reviewed for prescriptions for potentially inappropriate medications, urinary catheters, or physical restraints during the first 24 hours and the entire hospital stay. Medical records will be used to determine the total number of hospital acquired complications that may be related to CI; these include falls, injuries such as pulling out IV lines or urinary catheters, pressure ulcers, and new-onset delirium episodes that developed during hospitalization. Also, the time elapsed between screening for CI and the physician ordering a geriatric consultation will be calculated using the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Hospitalized in a medical ward
* Able to speak English
* Cognitive impairment based on screening at time of hospital admission

Exclusion Criteria:

* Previously enrolled in the study during prior hospitalization (for multiple admissions; only data from the first admission will be used)
* Enrolled in another clinical trial
* Does not have cognitive impairment based on screening at time of hospital admission

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 424 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Use of potentially inappropriate medications, urinary catheter or physical restraints, and length of time in initiating a referral order, as recorded in the electronic medical record | baseline and at discharge
Total number of hospital acquired complications recorded in the medical record that may be related to cognitive impairment (CI) | baseline and at discharge

SECONDARY OUTCOMES:
Length and cost of hospital stay from discharge records and billing system | baseline, at discharge, 6 months post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Malaz Boustani, MD, MPH, Principal Investigator — Regenstrief Institute, Inc.
Locations (1):
- Wishard Memorial Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Saravay SM, Kaplowitz M, Kurek J, Zeman D, Pollack S, Novik S, Knowlton S, Brendel M, Hoffman L. How do delirium and dementia increase length of stay of elderly general medical inpatients? Psychosomatics. 2004 May-Jun;45(3):235-42. doi: 10.1176/appi.psy.45.3.235. PMID 15123850
- [Background] Marcantonio ER, Goldman L, Mangione CM, Ludwig LE, Muraca B, Haslauer CM, Donaldson MC, Whittemore AD, Sugarbaker DJ, Poss R, et al. A clinical prediction rule for delirium after elective noncardiac surgery. JAMA. 1994 Jan 12;271(2):134-9. PMID 8264068
- [Background] Marcantonio ER, Juarez G, Goldman L, Mangione CM, Ludwig LE, Lind L, Katz N, Cook EF, Orav EJ, Lee TH. The relationship of postoperative delirium with psychoactive medications. JAMA. 1994 Nov 16;272(19):1518-22. PMID 7966844
- [Background] McCusker J, Cole MG, Dendukuri N, Belzile E. Does delirium increase hospital stay? J Am Geriatr Soc. 2003 Nov;51(11):1539-46. doi: 10.1046/j.1532-5415.2003.51509.x. PMID 14687382
- [Background] Marcantonio ER, Flacker JM, Michaels M, Resnick NM. Delirium is independently associated with poor functional recovery after hip fracture. J Am Geriatr Soc. 2000 Jun;48(6):618-24. doi: 10.1111/j.1532-5415.2000.tb04718.x. PMID 10855596
- [Background] Harwood DM, Hope T, Jacoby R. Cognitive impairment in medical inpatients. I: Screening for dementia--is history better than mental state? Age Ageing. 1997 Jan;26(1):31-5. doi: 10.1093/ageing/26.1.31. PMID 9143435